CLINICAL TRIAL: NCT00947557
Title: A Phase III, Randomized, Double-Blind, Placebo-controlled, Multicenter Study To Evaluate The Safety and Efficacy of Dutogliptin in Patients With Type 2 Diabetes Mellitus on Background Treatment With Glimepiride With or Without Metformin
Brief Title: Safety and Efficacy of Dutogliptin in Patients With Type 2 Diabetes Mellitus (T2DM) on Background Therapy With Glimepiride With or Without Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Phenomix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUT-MD-303
Record Dates: First submitted 2009-07-23; First posted 2009-07-28 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dutogliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dutogliptin (Active Comparator): Dutogliptin
  Interventions: Drug: Dutogliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutogliptin — Dutogliptin oral administration once daily on background of glimepiride with or without metformin
  Arms: Dutogliptin
Drug: Placebo — Placebo, oral administration once daily on background of glimepiride with or without metformin
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of dutogliptin in patients with type 2 diabetes mellitus (T2DM) who are receiving background therapy of glimepiride with or without metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed at least 3 months prior to Screening (Visit 1)
* BMI 20 to 48 kg/m2, inclusive
* HbA1c 7.0% - 10.0%, inclusive
* Age 18 to 85 years, inclusive

Exclusion Criteria:

* Currently on 3 or more oral antidiabetic drugs or insulin.
* Type 1 diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | HbA1c is drawn at Visit 1 (Week -16 to -4), Visit 3 (Week -2), Visit 4 (Week 0), Visit 5 (Week 4), Visit 6 (Week 10), Visit 7 (Week 18), Visit 8 (Week 26).

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG) | FPG is drawn at Visit 1 (Week -16 to -4), Visit 2 (Week -4), Visit 3 (Week -2), Visit 4 (Week 0), Visit 5 (Week 4), Visit 6 (Week 10), Visit 7 (Week 18), Visit 8 (Week 26).

CONTACTS AND LOCATIONS:
Overall Officials: Kaity Posada, PharmD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (147):
- United States (98):
  - Forest Investigative Site 064, Birmingham, Alabama
  - Forest Investigative Site 020, Birmingham, Alabama
  - Forest Investigative Site 025, Muscle Shoals, Alabama
  - Forest Investigative Site 059, Chandler, Arizona
  - Forest Investigative Site 113, Gilbert, Arizona
  - Forest Investigative Site 096, Litchfield, Arizona
  - Forest Investigative Site 080, Peoria, Arizona
  - Forest Investigative Site 098, Phoenix, Arizona
  - Forest Investigative Site 044, Scottsdale, Arizona
  - Forest Investigative Site 061, Anaheim, California
  - Forest Investigative Site 041, Chula Vista, California
  - Forest Investigative Site 049, Encinitas, California
  - Forest Investigative Site 022, Greenbrae, California
  - Forest Investigative Site 047, Harbor City, California
  - Forest Investigative Site 010, Huntington Park, California
  - Forest Investigative Site 070, Los Angeles, California
  - Forest Investigative Site 111, Northridge, California
  - Forest Investigative Site 031, Riverside, California
  - Forest Investigative Site 091, Roseville, California
  - Forest Investigative Site 067, Sacramento, California
  - Forest Investigative Site 112, Santa Ana, California
  - Forest Investigative Site 011, Walnut Creek, California
  - Forest Investigative Site 063, West Hills, California
  - Forest Investigative Site 088, Denver, Colorado
  - Forest Investigative Site 156, Boca Raton, Florida
  - Forest Investigative Site 004, Daytona Beach, Florida
  - Forest Investigative Site 052, DeLand, Florida
  - Forest Investigative Site 129, Hollywood, Florida
  - Forest Investigative Site 062, Jacksonville, Florida
  - Forest Investigative Site 050, Miami, Florida
  - Forest Investigative Site 021, Miami, Florida
  - Forest Investigative Site 122, Miami, Florida
  - Forest Investigative Site 125, Miami Lakes, Florida
  - Forest Investigative Site 069, New Port Richey, Florida
  - Forest Investigative Site 012, Ocala, Florida
  - Forest Investigative Site 015, Orlando, Florida
  - Forest Investigative Site 131, Ormond Beach, Florida
  - Forest Investigative Site 127, Pembroke Pines, Florida
  - Forest Investigative Site 018, Sarasota, Florida
  - Forest Investigative Site 075, St. Petersburg, Florida
  - Forest Investigative Site 026, West Palm Beach, Florida
  - Forest Investigative Site 045, Atlanta, Georgia
  - Forest Investigative Site 079, Augusta, Georgia
  - Forest Investigative Site 084, Roswell, Georgia
  - Forest Investigative Site 132, Roswell, Georgia
  - Forest Investigative Site 009, Meridian, Idaho
  - Forest Investigative Site 030, Peoria, Illinois
  - Forest Investigative Site 100, Evansville, Indiana
  - Forest Investigative Site 097, Evansville, Indiana
  - Forest Investigative Site 053, Kansas City, Kansas
  - Forest Investigative Site 008, Wichita, Kansas
  - Forest Investigative Site 107, Lexington, Kentucky
  - Forest Investigative Site 034, Covington, Louisiana
  - Forest Investigative Site 035, Baltimore, Maryland
  - Forest Investigative Site 046, Oxon Hill, Maryland
  - Forest Investigative Site 003, Brockton, Massachusetts
  - Forest Investigative Site 055, Brockton, Massachusetts
  - Forest Investigative Site 118, New Bedford, Massachusetts
  - Forest Investigative Site 007, Waltham, Massachusetts
  - Forest Investigative Site 002, Dearborn, Michigan
  - Forest Investigative Site 029, Saint Clair Shores, Michigan
  - Forest Investigative Site 054, Edina, Minnesota
  - Forest Investigative Site 072, Las Vegas, Nevada
  - Forest Investigative Site 065, Las Vegas, Nevada
  - Forest Investigative Site 101, Albuquerque, New Mexico
  - Forest Investigative Site 081, New Hyde Park, New York
  - Forest Investigative Site 016, New York, New York
  - Forest Investigative Site 094, Charlotte, North Carolina
  - Forest Investigative Site 051, Charlotte, North Carolina
  - Forest Investigative Site 058, Lenoir, North Carolina
  - Forest Investigative Site 038, Morehead City, North Carolina
  - Forest Investigative Site 040, Salisbury, North Carolina
  - Forest Investigative Site 082, Winston-Salem, North Carolina
  - Forest Investigative Site 039, Akron, Ohio
  - Forest Investigative Site 023, Cincinnati, Ohio
  - Forest Investigative Site 043, Columbus, Ohio
  - Forest Investigative Site 057, Dayton, Ohio
  - Forest Investigative Site 032, Kettering, Ohio
  - Forest Investigative Site 083, Bethany, Oklahoma
  - Forest Investigative Site 005, Eugene, Oregon
  - Forest Investigative Site 001, Medford, Oregon
  - Forest Investigative Site 126, Jenkintown, Pennsylvania
  - Forest Investigative Site 066, Philadelphia, Pennsylvania
  - Forest Investigative Site 036, Tipton, Pennsylvania
  - Forest Investigative Site 103, Greer, South Carolina
  - Forest Investigative Site 033, Pelzer, South Carolina
  - Forest Investigative Site 114, Chattanooga, Tennessee
  - Forest Investigative Site 104, Chattanooga, Tennessee
  - Forest Investigative Site 099, Arlington, Texas
  - Forest Investigative Site 056, Corpus Christi, Texas
  - Forest Investigative Site 071, Dallas, Texas
  - Forest Investigative Site 017, Dallas, Texas
  - Forest Investigative Site 014, Irving, Texas
  - Forest Investigative Site 109, San Antonio, Texas
  - Forest Investigative Site 119, San Antonio, Texas
  - Forest Investigative Site 076, Salt Lake City, Utah
  - Forest Investigative Site 028, Virginia Beach, Virginia
  - Forest Investigative Site 068, Renton, Washington
- Belarus (5):
  - Forest Investigative Site 208, Grodno, Belarus
  - Forest Investigative Site 202, Homyel, Belarus
  - Forest Investigative Site 207, Minsk, Belarus
  - Forest Investigative Site 209, Mogilev, Belarus
  - Forest Investigative Site 206, Vitebsk, Belarus
- Forest Investigative Site 302, Medellín, Antioquia, Colombia
- Hungary (2):
  - Forest Investigative Site 506, Budapest, Hungary
  - Forest Investigative Site 504, Szentes, Hungary
- India (18):
  - Forest Investigative Site 621, Hyderabad, Andhra Pradesh
  - Forest Investigative Site 614, Vijayawada, Andhra Pradesh
  - Forest Investigative Site 610, Visakhapatanam, Andhra Pradesh
  - Forest Investigative Site 609, Mapusa, Goa
  - Forest Investigative Site 618, Ahmedabad, Gujarat
  - Forest Investigative Site 620, Haryāna, Karnal
  - Forest Investigative Site 607, Bangalore, Karnataka
  - Forest Investigative Site 606, Bangalore, Karnataka
  - Forest Investigative Site 602, Bangalore, Karnataka
  - Forest Investigative Site 604, Bangalore, Karnataka
  - Forest Investigative Site 601, Mangalore, Karnataka
  - Forest Investigative Site 619, Palakkad, Kerala
  - Forest Investigative Site 616, Nagpur, Maharashtra
  - Forest Investigative Site 617, Nashik, Maharashtra
  - Forest Investigative Site 612, Pune, Maharashtra
  - Forest Investigative Site 603, Channi, Tamil Nadu
  - Forest Investigative Site 613, Chennai, Tamil Nadu
  - Forest Investigative Site 615, Vellore, Tamil Nadu
- Lithuania (5):
  - Forest Investigative Site 702, Kaunas, Lithuania
  - Forest Investigative Site 703, Kaunas, Lithuania
  - Forest Investigative Site 701, Kaunas, Lithuania
  - Forest Investigative Site 704, Klaipėda, Lithuania
  - Forest Investigative Site 705, Vilnius, Lithuania
- Peru (11):
  - Forest Investigative Site 804, Arequipa, Arequipa
  - Forest Investigative Site 803, Arequipa, Arequipa
  - Forest Investigative Site 812, Trujillo, La Libertad
  - Forest Investigative Site 811, Chiclayo, Lambayeque
  - Forest Investigative Site 805, Lima, Lima Province
  - Forest Investigative Site 813, Lima, Lima Province
  - Forest Investigative Site 801, Lima, Lima Province
  - Forest Investigative Site 807, Lima, Lima Province
  - Forest Investigative Site 809, Lima, Lima Province
  - Forest Investigative Site 808, Lima, Lima Province
  - Forest Investigative Site 802, Piura, Piura
- Romania (7):
  - Forest Investigative Site 909, Bacau, Romania
  - Forest Investigative Site 906, Bucharest, Romania
  - Forest Investigative Site 908, Bucharest, Romania
  - Forest Investigative Site 903, Satu Mare, Romania
  - Forest Investigative Site 901, Sibiu, Romania
  - Forest Investigative Site 905, Tg Mures, Romania
  - Forest Investigative Site 902, Timișoara, Romania